CLINICAL TRIAL: NCT03113578
Title: First-in-Human, Single Center, Evaluation of the DiLumen Device in Routine Colonoscopy
Brief Title: Evaluation of the DiLumen Device During Colonoscopy
Status: Completed | Type: Observational
Sponsor: Lumendi, LLC (Industry)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Reem Sharaiha, Assistant Professor of Medicine, Primary Investigator, Weill Medical College of Cornell University
Other Study IDs: DD-009; 1610017641 (Other: Weill-Cornell IRB)
Record Dates: First submitted 2017-03-15; First posted 2017-04-13 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Colon Polyp
Keywords: Balloon enteroscopy; colonoscopy; polyps
MeSH Terms: conditions — Colonic Polyps; Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: DiLumen — The study device is placed over a compatible endoscope to facilitate endoscopic diagnosis and treatment of any large intestine pathology with the use of double balloons
  Other Names: Endolumenal Interventional Platform

SUMMARY:
This is an observational registry study collecting data on the clinical performance of the study device (DiLumen™ ) for its intended use. The primary objective is to evaluate functional outcomes of the DiLumen device in humans. The secondary objective is to evaluate safety characteristics of the DiLumen device.

DETAILED DESCRIPTION:
The DiLumen™ Endolumenal Interventional Platform is a non-sterile, single-use, close-fitting sleeve that fits securely over a standard endoscope to stabilize it in the large intestine, and facilitates use of the endoscope for optical visualization, diagnosis, and treatment. It was developed by MINT (Minimally Invasive New Technology) at Weill Cornell. The technology has been licensed to Lumendi for commercialization.

The DiLumen Endolumenal Interventional Platform ("DiLumen" or "the device") is an accessory to an endoscope. The DiLumen dual balloon accessory is intended for use with any standard endoscope that has a distal tip outer diameter of 12.5 - 14.3 mm and a working length of 1680 mm or greater. The device is indicated to ensure complete positioning of an endoscope in the large intestine and assist with optical visualization, diagnosis, and endoscopic treatment.

The device received 510k clearance on Dec 6, 2016. The device is fully disposable, and consists of six major components that form its primary mechanical structure: (1) Fore Balloon; (2) Aft Balloon; (3) Sleeve; (4) Base; (5) Push Rod Mechanism; and (6) Inflation System.

The DiLumen utilizes two balloons to position and stabilize the endoscope within a patient's large intestine. After the device is installed over the endoscope, the endoscope/DiLumen are navigated to the target zone with the balloons deflated. The first balloon, the Aft balloon, is attached to the DiLumen sleeve. Once the clinician is at the target site, the Aft Balloon will be inflated until it contacts the intestinal wall near the proximal end of the articulating section of an endoscope. The second balloon, the Fore Balloon, is also attached to the sleeve via two flexible extension Push Rods and is deployed at the distal end of the endoscope at a variable distance. Once extended and inflated, the Fore Balloon contacts the patient's intestinal wall, and in combination with the Aft Balloon, creates an isolated diagnostic or therapeutic zone within a patient's large intestine. Both balloons are inflated or deflated with ambient air independently using an Inflation Handle with a squeeze bulb. The balloons assist with accessing and visualization of lesions behind folds and turns in the intestine, stabilizing the endoscope distal tip and establishing a Therapeutic Zone (TZ). Required insufflation within the therapeutic zone is minimized compared to typical colorectal endoscopic procedures, because the balloons enclose only a small portion (approximately 23 cm) of the large intestine.

The balloons and sleeve are designed to permit the usage of any standard endoscopic tool (such as biopsy forceps, snare, needle, etc.) through the endoscope working channel. The endoscope flexibility, maneuverability and functionalities (such as visualization, suction, insufflations, etc.) are unaffected by the presence of the DiLumen.

ELIGIBILITY:
Inclusion Criteria:

* Patients listed for routine surveillance colonoscopy for colorectal cancer and capable of giving informed consent

Exclusion Criteria:

* No patients less than 18 years of age.
* Any contraindication to routine surveillance colonoscopy
* History of open or laparoscopic colorectal surgery
* History of Inflammatory Bowel Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients listed for routine surveillance colonoscopy for colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Performance | Duration of procedure
  Ability to reach cecum with the study device and scope [Y or N]

SECONDARY OUTCOMES:
Incidence of Treatment Related Adverse Events | Up to 3 months
  No unintended visible mucosal injury on Dilumen withdrawal (above what is normally expected from colonoscopy)
Performance | Duration of Procedure
  Ability to inflate balloons in right colon and sigmoid colon and create a therapeutic zone [Y or N]

CONTACTS AND LOCATIONS:
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No